CLINICAL TRIAL: NCT00911066
Title: An Open-Label, Dose Escalation, Phase 1 Study of MLN4924, a Novel Inhibitor of Nedd8-Activating Enzyme, in Adult Patients With Acute Myelogenous Leukemia,Myelodysplastic Syndrome, and Acute Lymphoblastic Leukemia
Brief Title: MLN4924 for the Treatment of Acute Myelogenous Leukemia, Myelodysplastic Syndrome, and Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C15003
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes | interventions — pevonedistat; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MLN4924 (Experimental)
  Interventions: Drug: MLN4924
- Azacitidine (Experimental)
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: MLN4924 — MLN4924 intravenous (IV) on a 21-day cycle on one of the following schedules:
  * Days 1, 3, and 5, followed by a rest period of 16 days (Schedule A)
  * Days 1, 4, 8, and 11, followed by a rest period of 10 days (Schedule B)
  * Continuous weekly dosing on Days 1, 8, and 15 (Schedule C)
  * Days 1, 4, 11, 15 for Cycle 1 only; Days 1, 4, 8, 11 for all subsequent cycles (Schedule D)
  * Dosing on Days 1, 3, and 5 in patients with high-grade MDS or AML (Schedule E)
  Arms: MLN4924
Drug: Azacitidine — Azacitidine will be administered (IV or subcutaneous (SC)) on Days 8 to 12 and Days 15 and 16 in Cycle 1, and on Days 1 to 5 and Days 8 to 9 (Schedule D)
  Arms: Azacitidine

SUMMARY:
An open-label, multicenter, phase 1, dose escalation study of MLN4924 in adult patients with acute myelogenous leukemia (AML), high-grade myelodysplastic syndrome (MDS). The patient population will consist of adults previously diagnosed with AML including high-grade MDS for which standard curative, life-prolonging treatment does not exist or is no longer effective.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Have the following diagnosis:

  * AML or ALL (for the dose escalation phase only)including leukemia secondary to prior chemotherapy or resulting from an antecedent hematologic disorder, who have failed to achieve complete response (CR) or who have relapsed after prior therapy and are not candidates for potentially curative treatment.
  * Acute Promyelocytic Leukemia (APL) patients are not eligible
  * AML or ALL patients who are over age 60 and have not received prior therapy are also eligible if they are not candidates for standard induction chemotherapy
  * High-grade MDS, defined as > 10% blasts on bone marrow examination
  * Low-grade MDS, defined as < 10% blasts on bone marrow examination (Schedule B expansion cohort only)
* Patients who are willing to refrain from donating blood for at least 90 days after their final dose of MLN4924 and (for male patients) willing to refrain from donating semen for at least 4 months after their final dose of MLN4924
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Female patients who are postmenopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse
* Male patients who agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse
* Voluntary written consent
* Suitable venous access
* Adequate clinical laboratory values during the screening period as specified in the protocol
* Patients who are on hydroxyurea may be included in the study and may continue on hydroxyurea while participating in this study.

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Any serious medical or psychiatric illness
* Treatment with any investigational products
* Systemic antineoplastic therapy or radiotherapy within 14 days before the first dose of study drug, except for hydroxyurea
* Major surgery within 14 days before the first dose of study drug
* Life-threatening illness unrelated to cancer
* Clinically uncontrolled central nervous system (CNS) involvement
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
* Evidence of uncontrolled cardiovascular conditions as specified in the protocol
* Diarrhea > Grade 1, based on the NCI CTCAE categorization
* Systemic treatment with prohibited medications
* Ongoing anticoagulant therapy (eg, aspirin, Coumadin, heparin) that cannot be held to permit bone marrow sampling
* Use of acetaminophen, acetaminophen-containing products, and statins are not permitted on the day before dosing, day of dosing, and day after dosing with MLN4924

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-06; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Adverse events, serious adverse events, assessments of clinical laboratory values, and vital sign measurements | 12 months

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 12 months
Pharmacodynamic effects | 12 months
Assess disease response | 12 months
Heart corrected QT intervals | During screening and during Cycle 1, Days 1 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Stanford University Medical Center, Stanford, California
  - Robert H. Lurie Comprehensive Cancer Center Northwestern University, Chicago, Illinois
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Institute for Drug Development, San Antonio, Texas

REFERENCES:
- [Derived] Faessel HM, Mould DR, Zhou X, Faller DV, Sedarati F, Venkatakrishnan K. Population pharmacokinetics of pevonedistat alone or in combination with standard of care in patients with solid tumours or haematological malignancies. Br J Clin Pharmacol. 2019 Nov;85(11):2568-2579. doi: 10.1111/bcp.14078. Epub 2019 Sep 4. PMID 31355467
- [Derived] Swords RT, Erba HP, DeAngelo DJ, Bixby DL, Altman JK, Maris M, Hua Z, Blakemore SJ, Faessel H, Sedarati F, Dezube BJ, Giles FJ, Medeiros BC. Pevonedistat (MLN4924), a First-in-Class NEDD8-activating enzyme inhibitor, in patients with acute myeloid leukaemia and myelodysplastic syndromes: a phase 1 study. Br J Haematol. 2015 May;169(4):534-43. doi: 10.1111/bjh.13323. Epub 2015 Mar 2. PMID 25733005